CLINICAL TRIAL: NCT05870735
Title: The Patient Voice in Narcolepsy Clinical Trials: Reflections on Experiences and Outcomes
Brief Title: Discovering Factors in Narcolepsy Patients' Clinical Research Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 90685891
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Narcolepsy
Keywords: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational trial can provide a platform for patients to share experiences and perspectives on living with narcolepsy, which can inform the development of new treatments and support programs.

Overall, an observational clinical trial is an important tool for advancing the understanding of narcolepsy and improving outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is able and willing to comply with the treatment/follow-up schedule and requirements
* Patient must provide written informed consent

Exclusion Criteria:

* Women who are pregnant, intend to become pregnant, or are lactating
* Inability to perform regular electronic reporting
* Participants who are vulnerable to any intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational narcolepsy trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a narcolepsy clinical study. | 3 months
Number of narcolepsy study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fietze I, Bassetti CLA, Mayleben DW, Pain S, Seboek Kinter D, McCall WV. Efficacy and Safety of Daridorexant in Older and Younger Adults with Insomnia Disorder: A Secondary Analysis of a Randomised Placebo-Controlled Trial. Drugs Aging. 2022 Oct;39(10):795-810. doi: 10.1007/s40266-022-00977-4. Epub 2022 Sep 13. PMID 36098936
- [Background] Bassetti CLA, Adamantidis A, Burdakov D, Han F, Gay S, Kallweit U, Khatami R, Koning F, Kornum BR, Lammers GJ, Liblau RS, Luppi PH, Mayer G, Pollmacher T, Sakurai T, Sallusto F, Scammell TE, Tafti M, Dauvilliers Y. Narcolepsy - clinical spectrum, aetiopathophysiology, diagnosis and treatment. Nat Rev Neurol. 2019 Sep;15(9):519-539. doi: 10.1038/s41582-019-0226-9. Epub 2019 Jul 19. PMID 31324898
- [Background] Leschziner G. Narcolepsy: a clinical review. Pract Neurol. 2014 Oct;14(5):323-31. doi: 10.1136/practneurol-2014-000837. Epub 2014 May 15. PMID 24830461

DOCUMENTS (1):
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT05870735/ICF_000.pdf